CLINICAL TRIAL: NCT00153608
Title: Phase II Study of WT1 126-134 Peptide Vaccination in Combination With Adjuvants GM-CSF and KLH in Carcinomas
Brief Title: WT1 Peptid Vaccination in Carcinomas
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HaemaCBFWT104; EU
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2006-02-14 (Estimated); Status verified 2005-09

CONDITIONS: WT1 Expressing Carcinoma

INTERVENTIONS:
Biological: WT1 126-134 peptide

SUMMARY:
In this trial HLA-A2+ patients with WT1 expressing carcinomas are vaccinated with a peptide from the leukemia associated antigen WT1 together with immunological adjuvants KLH as T-helper protein and GM-CSF

ELIGIBILITY:
Inclusion Criteria:

* Metastatic cancer, no standard treatment option
* Resected cancer with minimal residual disease, no standard treatment option
* WT-1 expression
* HLA-A2

Exclusion Criteria:

* Concurrent chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25
Dates: Start 2004-04

PRIMARY OUTCOMES:
Clinical efficacy

SECONDARY OUTCOMES:
Immune response
Safety

CONTACTS AND LOCATIONS:
Overall Officials: Ulrich Keilholz, MD, Principal Investigator — Charité CBF
Locations (1):
- Hem&Onc Charité CBF, Berlin, Germany

REFERENCES:
- [Background] Keilholz U, Menssen HD, Gaiger A, Menke A, Oji Y, Oka Y, Scheibenbogen C, Stauss H, Thiel E, Sugiyama H. Wilms' tumour gene 1 (WT1) in human neoplasia. Leukemia. 2005 Aug;19(8):1318-23. doi: 10.1038/sj.leu.2403817. PMID 15920488